CLINICAL TRIAL: NCT04175873
Title: Effects of Music Therapy on Glutathione Peroxidase, Malondialdehyde and Pain in Oocyt Pick Up Patients: A Prospective, Randomized, Controlled Clinical Study)
Brief Title: The Effect of Music Therapy on Glutathione Peroxidase, Malondialdehyde and Pain in Oocyt Pick Up Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Yavuz Orak, Assistant Professor, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2019/14-09
Record Dates: First submitted 2019-10-30; First posted 2019-11-25 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Infertility; Anesthesia; Oxidative Stress; Pain, Postoperative
Keywords: music therapy; pain; oxidative stress
MeSH Terms: conditions — Infertility; Pain, Postoperative; Pain | interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: The patients will be listening to music with MP3 headphones for 1 hour preoperatively and throughout the operation.
Who Masked: Care Provider
Masking Description: The patients will be listening to music with MP3 headphones for 1 hour preoperatively and throughout the operation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group C (No Intervention): Control group.
- Group M (Experimental): Music group.Preoperative 1 hour and during the operation of Classical Turkish Music (Acemaşiran makam) listening group
  Interventions: Other: music

INTERVENTIONS:
Other: music — Patients will listen to music with MP3 headphones for 1 hour preoperatively and throughout the operation.
  Arms: Group M

SUMMARY:
It is used by music therapists to help the social, physical, emotional, psychological and psychological needs of patients. In a study, music has a positive effect on pain, anxiety, depression, shortness of breath, mood, facial expression and speech . The aim of this study was to investigate analgesia consumption during egg collection and postoperative period of music therapy and to compare and evaluate oxidative stress parameters in blood and follicle fluids.

DETAILED DESCRIPTION:
Patients will be divided into 2 groups. Group C (n = 30): Control group. Group M (n = 30): Music group. Preoperative 1 hour and during the operation of Classical Turkish Music (Acemaşiran makam) will listen to the group. After the patient is taken to the resting room, blood will be prepared for the operation (for malondialdehyde and glutathione peroxidase). Then STAI 1-2 anxiety form will be filled in under the supervision of the nurse. In Group M patients, blood will be taken to the patient resting room (for malondialdehyde, glutathione peroxidase). You will then play music with the MP3 headset for 1 hour. Then STAI 1-2 anxiety form will be filled in under the supervision of the nurse.Operation room will be taken. Remifentanil 0.5 mcg / kg and propofol 2 mg / kg will be administered for induction after all patients included in the study (Group C and Group M). Patients will be given BIS. Anesthetize BIS between 40-50. Hemodynamics follow-up (Systolic blood pressure, Diastolic blood pressure, Heart rate, Oxygen saturation) during the operation and the need for additional analgesia and anesthesia during the operation will be recorded. At the end of the operation, blood will be taken to compare the values of Oxidative Stress Parameters in the blood and follicle fluids. In the rest rooms, hemodynamics and pain follow-ups will be recorded at 1,5,15, 30, and 60 minutes. NRS (Numeric Rating Scale) will be used for pain monitoring. Analgesic needs of patients with pain will be met. Non-steroid anti-inflammatory (Naproxen Na) drug will be used for postoperative analgesia. At the end of the study, analgesia / anesthetic consumption, preoperative and postoperative blood oxidative stress parameters Glutathione peroxidase and Malondialdehyde will be compared in patients receiving music therapy and in patients without music therapy (control group). After the blood is drawn to both groups in the postoperative period, the STAI 1-2 questionnaire will be filled in under the supervision of the nurse and preoperative and postoperative comparisons will be made. The results will be correlated with the results.

Bispectral Index (BIS) monitoring is a new advanced electroencephalogram (EEG) based method for monitoring anesthetic depth (4). The monitor uses BIS analysis to obtain an index of anesthesia depth (5). BIS is a dimensionless number scaled from 100 to 0, and decreasing values show more sedation and hypnosis. A BIS value of 100 represents normal cortical electrical activity (an awake EEG), and a value of zero indicates a cortical electrical silence (cortical suppression).

ELIGIBILITY:
Inclusion Criteria:

* Patients with ASA 1
* Conscious patients
* Voluntary patients
* Patients without hearing problems
* Patients in the 18-35 age range
* Patients without music phobia will be included in the study
* Non-metabolic disease
* Patients without liver and kidney disease
* Patients without bleeding disorders

Exclusion Criteria:

* Non-volunteer
* Non-18-35 age range
* Patients without ASA 1
* Liver, Kidney and Metabolic Disease
* Unconscious
* Patients with hearing problems

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-11-25 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-05-15 (Actual)

PRIMARY OUTCOMES:
Glutathione Peroxidase markers with the music therapy | Change from baseline in one hour before operation and about 1st hour after operation
  To evaluate the impact on the circulating levels of Glutathione Peroxidase ü/ml,
Malondialdehyde markers with the music therapy | Change from baseline in one hour before operation and about 1st hour after operation
  To evaluate the impact on the circulating levels of Malondialdehyde nmol/ ml
Pain Score | after operation changing of pain level at 1 minute,5 minute,15 minute,30 minute, 60 minute
  VAS (Visual analog scale) Score. from 1 to 10 , 0: No pain, 10: 10 pain that can not be tolerated

SECONDARY OUTCOMES:
Hemodynamics | Changing during the operation, 1 minute, 3 minutes, 5 minutes, 7 minutes, 10 minutes, 15 minutes.Each unit will be evaluated separately within itself
  Systolic blood pressure (mmHg), diastolic blood pressure (mm Hg), mean arterial pressure (mmHg),
Hemodynamics | Changing after the operation in 1 minute, 5 minutes, 15 minutes, 30 minutes, 60 minutes.Each unit will be evaluated separately within itself
  Systolic blood pressure (mmHg), diastolic blood pressure (mmHg), mean arterial pressure (mmHg), heart rate,
Heart rate | Changing after the operation in 1 minute, 5 minutes, 15 minutes, 30 minutes, 60 minutes.Each unit will be evaluated separately within itself
  heart rate
STAI | Change from baseline in one hour before operation and about 1st hour after operation
  State-Trait Anxiety Inventory Score

CONTACTS AND LOCATIONS:
Overall Officials: yavuz orak, Principal Investigator — Kahramanmaraş Sutcu Imam University Faculty of Medicine
Locations (2):
- Turkey (Türkiye) (2):
  - Kahramanmaras Sutcu Imam Univercity Faculty of edicine, Kahramanmaraş, Onikişubat
  - Kahramanmaras Sutcu Imam University Faculty of Medicine, Kahramanmaraş, Onikişubat